CLINICAL TRIAL: NCT04425980
Title: The Efficacy of Two Models of Intensive Upper Limb Training On Quality of Life in Children With Hemiplegic Cerebral Palsy Attending Regular School in Mus Province: A Randomized Controlled Trial
Brief Title: The Efficacy of Two Models of Intensive Upper Limb Training on Quality of Life in Children With Congenital Hemiplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Hasan Bingöl, Academician (Lecturer, Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: no any sponsor
Record Dates: First submitted 2020-06-05; First posted 2020-06-11 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Hemiplegia; Congenital
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Intervention Model Description: a total of 30 children met inclusion criteria (grades 1-4) were randomly assigned to one of two groups (modified constraint-induced movement therapy or Bimanual training), at an equal number and probability
Who Masked: Participant
Masking Description: by concealing the other allocated intervention from participants / unaware of the presence of a second intervention approach
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Constraint-Induced Movement Therapy (test treatments) (Experimental): A list of fine and motor activities consisted of the functional tasks or play activities such as school-education and sports activities, manipulative games, arts, and crafts, etc. to elicit the maximum capacity of the more affected upper limb was created according to the procedure of modified constraint-induced movement therapy (Gordon et al., 2005) and Bimanual training. In addition, specific activities were also chosen in terms of deficit of interest, participant preference (on the condition of having potential effects on hand skills) and parent/guardian, or their teacher's request. In case of activities requiring both hand use, such as stabilizing paper during the painting or holding the bricks of lego on the ground, the treating physiotherapist undertook a role as a dominant hand
  Interventions: Other: Modified Constraint-Induced Movement Therapy
- Bimanual training (Active Comparator): For the Bimanual training, skilled, repetitive, and structured bimanual activities (part or whole task practice) were used to promote bimanual hand use and improve movement deficits determined before the intervention. All targeted deficits of interest were addressed within the context of the selected activity. Specifically, symmetrical bilateral movements were utilized to augment neural input from both sides. Also, meaningful activities such as buttoning and zipping-up trousers, etc. were used to ensure a transition from structured setting to real-life activities
  Interventions: Other: Modified Constraint-Induced Movement Therapy

INTERVENTIONS:
Other: Modified Constraint-Induced Movement Therapy — intensive use of more affected arm in structured setting

SUMMARY:
This study compared the effectiveness of two-mode of activity-based upper limb rehabilitation (Modified Constraint-Induced Movement Therapy and Bimanual training) on health-related quality of life outcomes in school-aged children with cerebral palsy

DETAILED DESCRIPTION:
A total of 52 primary schools were screened comprehensively to determine children conforming specifications of the inclusion criteria. Demographic characteristics (e.g. age, gender, affected side) and severity of functional impairment dealing with cognitive /communication, manual ability and mobility were noted. After a comprehensive screening, a total of 30 children met inclusion criteria (grades 1-4) were randomly assigned to one of two groups (Modified Constraint-Induced Movement Therapy or Bimanual training), at an equal number and probability. Children blinded to group allocation were delivered activity-based upper limb training in the context of Modified Constraint-Induced Movement Therapy or Bimanual training, at a similar dose and frequency (10 weeks/3 days per week/2.5 hours per day). 1 out of 3 sessions per week was carried out in the school time (during the art or physical education class), while 2 out of 3 sessions were carried out in rehabilitation centers which the children regularly attend for regular care 2-day weekly. All participating children continued to receive their standard care (90 minutes per week) throughout the study period.

During the 1-month screening period, physical characteristics of participants were described through classification systems including The Communication Function Classification System, The Manual Ability Classification System , and The Gross Motor Function Classification System. Participating children were evaluated before the study entry (T1), immediately postintervention (T2), and at 16 weeks postintervention (T3) using the KIDSCREEN-27 questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of congenital hemiplegia,
* Must be able to grasp objects

Exclusion Criteria:

* Cerebral palsy dependent severe emotional difficulties

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in quality of life on the 5 point KIDSCREEN-27 questionnaire at post intervention | From baeline to post-intervention, up to 16 weeks
  The KIDSCREEN instruments have been established to report various subdomains of QOL about physical, emotional, mental and social well-being in school-aged children and adolescents

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Bingöl, MSc, Principal Investigator — Muş Alparslan University; Mintaze Kerem Günel, PhD, Study Chair — Hacettepe University; Halil ALKAN, PhD, Principal Investigator — Muş Alparslan University
Locations (1):
- Mus Alparslan University, Muş, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No